CLINICAL TRIAL: NCT05381493
Title: Incidence and Outcomes of Acute Kidney Injury in Trauma Patients Admitted to Critical Care
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Bengi Şafak (Unknown); Keziban Sanem Çakar Turhan (Unknown); Mustafa Onur Karaca (Unknown); Uğur Aydoğan (Unknown); Ali Abbas Yılmaz (Unknown); Mustafa Kemal Bayar (Unknown)
Responsible Party: Principal Investigator, Süheyla Karadağ Erkoç, Anesthesiology and Reanimation, Ankara University
Other Study IDs: AnkaraUTraumaAKI
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury; Trauma; Complications
Keywords: Trauma; Acute Kidney Injury; Intensive Care Unit
MeSH Terms: conditions — Acute Kidney Injury; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication that increases lenght of stay and mortality in trauma patients admitted to the intensive care unit (ICU). The aim of this study is to identify the incidence and outcomes of trauma patients, defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria, at single center level 3 ICU.

DETAILED DESCRIPTION:
Trauma can cause high mortality and morbidity by affecting different organ systems. Acute kidney injury (AKI) is a common complication in trauma patients admitted to the intensive care unit (ICU). Direct kidney injury, hypotension, hypoperfusion, rhabdomyolysis, abdominal compartment syndrome, sepsis and critical care medications are possible causes of AKI in trauma patients. The incidence of AKI can be up to 10%, and mortality rate up to 60-80% in trauma patients. Since AKI is not only a rare complication but also a risk factor for mortality in critically ill trauma patients, it is essential to establish a strategy to prevent AKI and related complications, to determine the incidence and risk factors of AKI, and to improve patients outcomes. Survivors of AKI may have variable recovery of kidney function and might prone to late morbidity and mortality. In this study incidence of AKI was defined using the KDIGO criteria according to the change of serum creatine levels.

171 all type of trauma patients admitted to level 3 ICU, from January 2014 to December 2018 included the retrospectve observational study. Demographic data, type of injury, rates of complications, risk factors for AKI, mortality, lenght of stay (LOS) in ICU were evaluated. Acute Physiology and Chronic Health Evaluation (APACHE II and IV) score, Simplified Acute Physiology Score (SAPS II and III), Glasgow Coma Scale (GCS), Injury Severity Score (ISS) and, Trauma Injury Severity Score (TRISS) were calculated on the day of admission. AKI was defined using the KDIGO criteria according to the serum creatinine. The SPSS 11.5 program was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* all type of trauma patients admitted to level 3 ICU, from January 2014 to December 2018

Exclusion Criteria:

-

Ages: 18 Years to 97 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all type of trauma patients admitted to level 3 ICU
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury in trauma patients | one week
  Kidney Disease Improving Global Outcomes (KDIGO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Karadağ Erkoç, Principal Investigator — Ankara University
Locations (1):
- Süheyla Karadağ Erkoç, Ankara, Turkey (Türkiye)